CLINICAL TRIAL: NCT01521923
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Certolizumab Pegol in Combination With Methotrexate for Inducing and Sustaining Clinical Response in the Treatment of DMARD-Naïve Adults With Early Active Rheumatoid Arthritis
Brief Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Certolizumab Pegol in Combination With Methotrexate in the Treatment of Disease Modifying Antirheumatic Drugs (DMARD)-naïve Adults With Early Active Rheumatoid Arthritis
Acronym: C-early
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA0055 Period 2; 2011-001729-25 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2012-01-19; First posted 2012-01-31 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab Pegol - Cimzia; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CZP 200 mg Q2W + Methotrexate (Experimental)
  Interventions: Biological: Certolizumab Pegol + Methotrexate (MTX)
- CZP 200 mg Q4W + Methotrexate (Experimental)
  Interventions: Biological: Certolizumab Pegol + Methotrexate (MTX)
- Placebo + Methotrexate (Placebo Comparator)
  Interventions: Biological: Placebo + Methotrexate (MTX)

INTERVENTIONS:
Biological: Certolizumab Pegol + Methotrexate (MTX) — Prefilled syringes containing an injectable volume of 1 ml of solution for injection CZP for single use at dosage strength of 200 mg/ml.
  On a maintenance dose of 200 mg every 2 Weeks (Q2W) until Week 102. On a maintenance dose of 200 mg every 4 Weeks (Q4W) until Week 102/ Placebo (PBO) 1 syringe every 4 Weeks (Q4W).
  CZP and PBO administration to be staggered 2 Weeks apart to maintain blind.
  The MTX treatment is to remain between 15-25 mg/week.
  Other Names: Cimzia; CZP; MTX
  Arms: CZP 200 mg Q2W + Methotrexate; CZP 200 mg Q4W + Methotrexate
Biological: Placebo + Methotrexate (MTX) — 1 syringe of Placebo every 2 Weeks and MTX.
  The MTX treatment is to remain between 15-25 mg/week.
  Other Names: MTX
  Arms: Placebo + Methotrexate

SUMMARY:
This study is intended to evaluate the efficacy and safety of Certolizumab Pegol (CZP) in combination with Methotrexate (MTX) for sustaining clinical response achieved in study RA0055 Period 1 [NCT01519791]. Subjects entering this study RA0055 Period 2 achieved sustained Low Disease Activity at Week 52 in study RA0055 Period 1.

ELIGIBILITY:
Inclusion Criteria:

- Those subjects in previous study RA0055 Period 1 who are in sustained LDA (defined as DAS28[ESR] ≤ 3.2 at Weeks 40 and 52) at Week 52 in previous study RA0055 Period 1

Exclusion Criteria:

- Those subjects in previous study RA0055 Period 1 who are NOT in sustained LDA (defined as DAS28[ESR] ≤ 3.2 at Weeks 40 and 52) at Week 52 in previous study RA0055 Period 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (178):
- United States (70):
  - 209, Birmingham, Alabama
  - 170, Huntsville, Alabama
  - 180, Mobile, Alabama
  - 247, Glendale, Arizona
  - 165, Paradise Valley, Arizona
  - 234, Paradise Valley, Arizona
  - 243, Phoenix, Arizona
  - 251, Tucson, Arizona
  - 160, Covina, California
  - 257, Hemet, California
  - 159, Los Angeles, California
  - 201, San Leandro, California
  - 202, Upland, California
  - 172, Whittier, California
  - 190, Fort Lauderdale, Florida
  - 196, Jupiter, Florida
  - 238, Lake Mary, Florida
  - 232, Miami, Florida
  - 213, Naples, Florida
  - 214, Ocala, Florida
  - 237, Orange Park, Florida
  - 255, Orlando, Florida
  - 163, Palm Harbor, Florida
  - 166, Plantation, Florida
  - 192, Sarasota, Florida
  - 200, Vero Beach, Florida
  - 226, Coeur d'Alene, Idaho
  - 244, Springfield, Illinois
  - 224, South Bend, Indiana
  - 215, Cedar Rapids, Iowa
  - 191, Wichita, Kansas
  - 210, Wichita, Kansas
  - 177, Hagerstown, Maryland
  - 199, Kalamazoo, Michigan
  - 198, Eagan, Minnesota
  - 203, Tupelo, Mississippi
  - 179, St Louis, Missouri
  - 181, Lincoln, Nebraska
  - 256, Reno, Nevada
  - 229, Lebanon, New Hampshire
  - 228, Clifton, New Jersey
  - 207, Albuquerque, New Mexico
  - 176, Brooklyn, New York
  - 242, Plainview, New York
  - 227, Rochester, New York
  - 236, Durham, North Carolina
  - 245, Middleburg Heights, Ohio
  - 241, Oklahoma City, Oklahoma
  - 186, Portland, Oregon
  - 195, Bethlehem, Pennsylvania
  - 167, Duncansville, Pennsylvania
  - 168, Wyomissing, Pennsylvania
  - 189, Charleston, South Carolina
  - 205, Columbia, South Carolina
  - 204, Hendersonville, Tennessee
  - 217, Allen, Texas
  - 185, Amarillo, Texas
  - 161, Austin, Texas
  - 178, Corpus Christi, Texas
  - 162, Dallas, Texas
  - 184, Houston, Texas
  - 206, Houston, Texas
  - 223, Houston, Texas
  - 158, Mesquite, Texas
  - 175, Nassau Bay, Texas
  - 249, Plano, Texas
  - 197, San Antonio, Texas
  - 233, Kennewick, Washington
  - 183, Clarksburg, West Virginia
  - 174, Glendale, Wisconsin
- Argentina (4):
  - 276, Buenos Aires
  - 284, Rosario
  - 279, San Juan
  - 291, San Miguel de Tucumán
- Australia (8):
  - 6, Coffs Harbour, New South Wales
  - 2, Herson, Queensland
  - 1, Maroochydore, Queensland
  - 8, Woodville South, South Australia
  - 5, Fitzroy, Victoria
  - 4, Geelong, Victoria
  - 3, Malvern, Victoria
  - 7, Perth, Western Australia
- 50, Vienna, Austria
- Belgium (4):
  - 51, Brussels
  - 126, Gilly
  - 36, Kortrijk
  - 65, Yvoir
- Canada (4):
  - 240, Kelowna, British Columbia
  - 235, Hamilton, Ontario
  - 188, Montreal, Quebec
  - 194, Trois-Rivières, Quebec
- Colombia (8):
  - 303, Barranquilla
  - 272, Bogotá
  - 293, Bogotá
  - 299, Bogotá
  - 297, Bucaramanga
  - 288, Chía
  - 271, Medellín
  - 298, Medellín
- Czechia (4):
  - 108, Brno
  - 124, Bruntál
  - 38, Hradec Králové
  - 37, Prague
- France (5):
  - 16, Le Kremlin-Bicêtre
  - 85, Le Mans
  - 88, Montpellier
  - 34, Orléans
  - 79, Strasbourg
- Germany (16):
  - 52, Bad Doberan
  - 17, Bayreuth
  - 113, Berlin
  - 120, Berlin
  - 89, Erfurt
  - 70, Frankfurt
  - 71, Hamburg
  - 81, Hildesheim
  - 127, Lingen
  - 61, München
  - 53, Planegg
  - 132, Ratingen
  - 49, Rendsburg
  - 69, Rheine
  - 114, Würzburg
  - 59, Zerbst
- Hungary (6):
  - 18, Budapest
  - 21, Budapest
  - 86, Eger
  - 131, Szolnok
  - 110, Szombathely
  - 19, Veszprém
- Ireland (3):
  - 33, Cork
  - 54, Dublin
  - 32, Limerick
- Italy (5):
  - 115, Ferrara
  - 122, Milan
  - 40, Reggio Emilia
  - 72, Roma
  - 41, Verona
- Mexico (6):
  - 281, Durango
  - 286, Guadalajara
  - 292, Mexico City
  - 302, Mérida
  - 280, Monterrey
  - 294, San Luis Potosí City
- 78, Monaco, Monaco
- 42, Leiden, Netherlands
- Poland (7):
  - 128, Bydgoszcz
  - 67, Elblag
  - 99, Krakow
  - 92, Poznan
  - 74, Torun
  - 100, Warsaw
  - 44, Wroclaw
- Romania (7):
  - 58, Brasov
  - 111, Bucharest
  - 22, Bucharest
  - 25, Bucharest
  - 26, Bucharest
  - 24, Iași
  - 57, LASI
- Spain (3):
  - 93, A Coruña
  - 47, Madrid
  - 63, Santiago de Compostela
- Sweden (6):
  - 76, Gothenburg
  - 82, Huddinge
  - 106, Lund
  - 123, Malmo
  - 77, Stockholm
  - 75, Uppsala
- Switzerland (2):
  - 118, Fribourg
  - 68, Sankt Gallen
- United Kingdom (7):
  - 125, Cannock
  - 105, Dudley
  - 56, Leeds
  - 121, London
  - 27, London
  - 80, Sheffield
  - 119, York

REFERENCES:
- [Result] Emery P, Bingham CO 3rd, Burmester GR, Bykerk VP, Furst DE, Mariette X, van der Heijde D, van Vollenhoven R, Arendt C, Mountian I, Purcaru O, Tatla D, VanLunen B, Weinblatt ME. Certolizumab pegol in combination with dose-optimised methotrexate in DMARD-naive patients with early, active rheumatoid arthritis with poor prognostic factors: 1-year results from C-EARLY, a randomised, double-blind, placebo-controlled phase III study. Ann Rheum Dis. 2017 Jan;76(1):96-104. doi: 10.1136/annrheumdis-2015-209057. Epub 2016 May 10. PMID 27165179
- [Result] Weinblatt ME, Bingham CO 3rd, Burmester GR, Bykerk VP, Furst DE, Mariette X, van der Heijde D, van Vollenhoven R, VanLunen B, Ecoffet C, Cioffi C, Emery P. A Phase III Study Evaluating Continuation, Tapering, and Withdrawal of Certolizumab Pegol After One Year of Therapy in Patients With Early Rheumatoid Arthritis. Arthritis Rheumatol. 2017 Oct;69(10):1937-1948. doi: 10.1002/art.40196. Epub 2017 Sep 12. PMID 28666080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in January 2012.
Pre-assignment Details: Participant Flow refers to the Safety Set 2 (SS2) which consists of all subjects randomized into Period 1 who had received at least 1 dose of study medication (CZP/PBO) in Period 2. Of the 359 enrolled patients, 357 are included in the SS2.
Groups:
- PBO+MTX / PBO+MTX: Placebo (PBO) + Methotrexate (MTX) in Period 1
  1 syringe PBO every 2 Weeks + MTX in Period 2
- CZP+MTX / PBO+MTX: Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe PBO every 2 Weeks + MTX in Period 2
- CZP+MTX / CZP Q4W+MTX: Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe 200 mg Certolizumab pegol (CZP) every 4 Weeks/ 1 syringe Placebo (PBO) every 4 Weeks (CZP and PBO administration to be staggered 2 weeks apart to maintain blind) + MTX in Period 2
- CZP+MTX / CZP Q2W+MTX: Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe 200 mg Certolizumab pegol (CZP) every 2 Weeks + MTX in Period 2
Period: Overall Study
Arm/Group | PBO+MTX / PBO+MTX | CZP+MTX / PBO+MTX | CZP+MTX / CZP Q4W+MTX | CZP+MTX / CZP Q2W+MTX
Started | 66 | 81 | 127 | 83
Completed | 59 | 72 | 112 | 70
Not Completed | 7 | 9 | 15 | 13
Not completed — AE, serious fatal | 1 | 0 | 0 | 0
Not completed — SAE, non-fatal | 0 | 2 | 2 | 0
Not completed — AE, non-serious, non-fatal | 1 | 3 | 6 | 2
Not completed — SAE, nonfatal + AE, non-serious nonfatal | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2
Not completed — Other | 2 | 1 | 3 | 6
Not completed — AE, captured in Period 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline refers to Baseline from Period 1. Only subjects who entered Period 2 are included. Characteristics refer to the Safety Set 2 (SS2).
Groups:
- PBO+MTX / PBO+MTX: Placebo (PBO) + Methotrexate (MTX) in Period 11 syringe PBO every 2 Weeks + MTX in Period 2
- CZP+MTX / PBO+MTX: Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 11 syringe PBO every 2 Weeks + MTX in Period 2
- CZP+MTX / CZP Q4W+MTX: Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 11 syringe 200 mg Certolizumab pegol (CZP) every 4 Weeks/ 1 syringe Placebo (PBO) every 4 Weeks (CZP and PBO administration to be staggered 2 weeks apart to maintain blind) + MTX in Period 2
- CZP+MTX / CZP Q2W+MTX: Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 11 syringe 200 mg Certolizumab pegol (CZP) every 2 Weeks + MTX in Period 2
Arm/Group | PBO+MTX / PBO+MTX | CZP+MTX / PBO+MTX | CZP+MTX / CZP Q4W+MTX | CZP+MTX / CZP Q2W+MTX | Total Title
Number analyzed (Participants) | 66 | 81 | 127 | 83 | 357
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 0 | 2
  Between 18 and 65 years | 54 | 70 | 114 | 72 | 310
  >=65 years | 12 | 11 | 11 | 11 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.7) | 47.9 (14.1) | 49.1 (12.5) | 49.1 (13.2) | 49.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 59 | 87 | 65 | 265
  Male | 12 | 22 | 40 | 18 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) <= 3.2 at Week 104 in RA0055 Period 2 Without Flaring
Description: This Outcome Measure includes all subjects that have a DAS28 [ESR] <= 3.2 from the start of RA0055 Period 2 (Week 52 of RA0055 Period 1) to Week 104 in RA0055 Period 2 without flaring.
Time Frame: Week 104 in RA0055 Period 2
Population: FAS2 with NRI. FAS2 did not include subjects who had received PBO+MTX in Period 1 as this was not part of the study objectives for the Period 2 efficacy analyses
  1 subject in the CZP+MTX/CZP Q2W+MTX and 1 in the CZP+MTX/PBO+MTX arm had post Week 52 assessments, but weren´t dosed in Period 2. They are included in the FAS2, but excluded from the SS2
Measure: Number; unit: percentage of subjects
Groups:
- CZP+MTX / PBO+MTX (Full Analysis Set [FAS]): Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe PBO every 2 Weeks + MTX in Period 2
- CZP+MTX / CZP Q4W+MTX (Full Analysis Set): Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe 200 mg Certolizumab pegol (CZP) every 4 Weeks/ 1 syringe Placebo (PBO) every 4 Weeks (CZP and PBO administration to be staggered 2 weeks apart to maintain blind) + MTX in Period 2
- CZP+MTX / CZP Q2W+MTX (Full Analysis Set): Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe 200 mg Certolizumab pegol (CZP) every 2 Weeks + MTX in Period 2
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set [FAS]) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 39.2 | 53.2 | 48.8
Statistical Analysis 1: Comparison: CZP+MTX / PBO+MTX (Full Analysis Set [FAS]) vs CZP+MTX / CZP Q2W+MTX (Full Analysis Set); In order to control the overall study-wise Type I error rate at 5 %, hypothesis testing was performed in a hierarchical order beginning with the CZP standard maintenance dosing (200 mg Q2W) + MTX group vs the CZP stopped dosing (PBO) + MTX group. If this analysis was statistically significant at the alpha =0.05 level, then an additional comparison of the CZP reduced frequency dosing (200 mg Q4W) + MTX group vs the CZP stopped dosing + MTX group was performed with testing at the alpha =0.05 level; Test type: Superiority or Other; p = 0.112, Regression, Logistic; Odds Ratio (OR) = 1.719, 95% CI 2-sided [0.881 to 3.354]
Statistical Analysis 2: Comparison: CZP+MTX / PBO+MTX (Full Analysis Set [FAS]) vs CZP+MTX / CZP Q4W+MTX (Full Analysis Set); In order to control the overall study-wise Type I error rate at 5 %, hypothesis testing was performed in a hierarchical order. A hierarchical test procedure was applied to protect the Overall significance level for the multiplicity of endpoints. Hypothesis testing was performed in the following predefined order, each at a 2-sided 95 % alpha level; Test type: Superiority or Other; p = 0.041, Regression, Logistic; Odds Ratio (OR) = 1.889, 95% CI 2-sided [1.026 to 3.480]

2. Secondary Outcome: Percentage of Subjects With Disease Activity Score 28 [ESR] (DAS28 [ESR]) < 2.6 at Week 52 in Previous Study RA0055 Period 1 Who Maintain a DAS28 [ESR] < 2.6 From Week 52 in RA0055 Period 1 Through Week 104 in RA0055 Period 2 Without Flaring
Description: DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x PtGADA, where 28 joints are examined and a lower score indicates less disease activity.
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: Full Analysis Set Period 2 (FAS2) with Non-Responder Imputation (NRI). FAS2 did not include subjects who had received PBO + MTX in Period 1 as this was not part of the study objectives for the Period 2 efficacy analyses.
Measure: Number; unit: percentage of subjects
Groups:
- CZP+MTX / PBO+MTX (Full Analysis Set): Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe PBO every 2 Weeks + MTX in Period 2
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 51 | 83 | 50
percentage of subjects | 33.3 | 43.4 | 44.0

3. Secondary Outcome: Change From Baseline in Previous Study RA0055 Period 1 in Modified Total Sharp Score (mTSS) to Week 104 in RA0055 Period 2
Description: Van der Heijde modified Total Sharp Score (mTSS) is a methodology to assess the degree of joint damage by quantifying the extent of bone erosions and joint space narrowing for 44 and 42 joints, respectively. The mTSS ranges from 0 to 448, with higher scores representing greater damage.
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: The Radiographic Set Period 2 (RAD2) consisted of those subjects in the FAS2 who had provided valid radiographs at Baseline, at Week 52, and at Week 104 or the Withdrawal Visit.
  RAD2 did not include subjects who had received PBO + MTX in Period 1 as this was not part of the study objectives for the Period 2 efficacy analyses.
Measure: Median (Full Range); unit: units on a scale
Groups:
- CZP+MTX / PBO+MTX (Radiographic Set): Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe PBO every 2 Weeks + MTX in Period 2
- CZP+MTX / CZP Q4W+MTX (Radiographic Set): Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe 200 mg Certolizumab pegol (CZP) every 4 Weeks/ 1 syringe Placebo (PBO) every 4 Weeks (CZP and PBO administration to be staggered 2 weeks apart to maintain blind) + MTX in Period 2
- CZP+MTX / CZP Q2W+MTX (Radiographic Set): Certolizumab pegol (CZP) 200 mg Q2W + Methotrexate (MTX) in Period 1
  1 syringe 200mg Certolizumab pegol (CZP) every 2 Weeks + MTX in Period 2
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
units on a scale | 0 [-5 to 28] | 0 [-9 to 9] | 0 [-2 to 9]

4. Secondary Outcome: Change From Week 52 in Previous Study RA0055 Period 1 in Modified Total Sharp Score (mTSS) to Week 104 in RA0055 Period 2
Description: as for outcome 3
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
units on a scale | 0 [-3 to 50] | 0 [-9 to 7] | 0 [-4 to 4]

5. Secondary Outcome: Percentage of Subjects With Radiographic Non-progression From Baseline in Previous Study RA0055 Period 1 to Week 104 in RA0055 Period 2
Description: Radiographic nonprogression is defined as change in modified Total Sharp Score (mTSS) <= 0.5.
  Van der Heijde modified Total Sharp Score (mTSS) is a methodology to assess the degree of joint damage by quantifying the extent of bone erosions and joint space narrowing for 44 and 42 joints, respectively. The mTSS ranges from 0 to 448, with higher scores representing greater damage.
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
percentage of subjects | 69.3 | 77.9 | 79.2

6. Secondary Outcome: Percentage of Subjects With Radiographic Non-progression From Week 52 in Previous Study RA0055 Period 1 to Week 104 in RA0055 Period 2
Description: as for outcome 5
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
percentage of subjects | 80.0 | 84.1 | 90.3

7. Secondary Outcome: Change From Baseline in Previous Study RA0055 Period 1 in the Joint Erosion Score to Week 104 in RA0055 Period 2
Description: Erosions were assessed in 16 locations per hand and 6 joints per foot. Erosions for each hand location were scored from 0 to 5, with 0 indicating no erosion. Scores 1 to 5 may have included combinations of discrete erosion(s) and/or large erosions. Erosions for each foot joint were scored from 0 to 10, with 0 indicating no erosions.
  The minimum possible total erosion score for all 32-hand joints was 0, the maximum possible erosion score for all 32-hand joints was 160. The minimum possible total erosion score for all 12-feet joints was 0, the maximum possible erosion score for all 12 feet joints was 120. Thus, the minimum possible total erosion score for hands and feet was 0, the maximum possible total erosion score for hands and feet was 280. Higher values represent greater damage.
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
units on a scale | 0 [-4 to 18] | 0 [-8 to 7] | 0 [-2 to 9]

8. Secondary Outcome: Change From Week 52 in Previous Study RA0055 Period 1 in the Joint Erosion Score to Week 104 in RA0055 Period 2
Description: as for outcome 7
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
units on a scale | 0 [-3 to 36] | 0 [-8 to 5] | 0 [-2 to 4]

9. Secondary Outcome: Change From Baseline in Previous Study RA0055 Period 1 in the Joint Narrowing Score to Week 104 in RA0055 Period 2
Description: Joint space narrowing (JSN) was assessed in 15 locations per hand and 6 locations per foot. Joint space narrowing for each location was scored from 0 to 4, with 0 indicating no narrowing. The minimum possible score for JSN in all 30 hand joints was 0, the maximum possible score for JSN in all 30 hand joints was 120. The minimum possible score for JSN in all 12 feet joints was 0, the maximum possible score for JSN in all 12 feet joints was 48. Thus, the minimum possible total JSN score for hands and feet was 0, the the maximum possible total JSN score for Hands and feet was 168. Higher values represent greater damage.
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
units on a scale | 0 [-3 to 12] | 0 [-4 to 4] | 0 [-2 to 2]

10. Secondary Outcome: Change From Week 52 in Previous Study RA0055 Period 1 in the Joint Narrowing Score to Week 104 in RA0055 Period 2
Description: as for outcome 9
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Radiographic Set) | CZP+MTX / CZP Q4W+MTX (Radiographic Set) | CZP+MTX / CZP Q2W+MTX (Radiographic Set)
Number analyzed (Participants) | 75 | 113 | 72
units on a scale | 0 [-2 to 14] | 0 [-3 to 5] | 0 [-4 to 2]

11. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 104 in RA0055 Period 2
Description: The assessments are based on a 20 % or greater improvement from Baseline in previous study RA0055 Period 1 in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 74.7 | 86.5 | 73.8

12. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 104 in RA0055 Period 2
Description: The assessments are based on a 50 % or greater improvement from Baseline in previous study RA0055 Period 1 in the number of tender joints, a 50 % or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 68.4 | 80.2 | 71.4

13. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 104 in RA0055 Period 2
Description: The assessments are based on a 70 % or greater improvement from Baseline in previous study RA0055 Period 1 in the number of tender joints, a 70 % or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 60.8 | 70.6 | 63.1

14. Secondary Outcome: Percentage of Subjects Meeting the 2011 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Remission Criteria at Week 104 in RA0055 Period 2
Description: The ACR/EULAR 2011 remission criteria is defined as:
  Tender Joint Count (TJC) <= 1, Swollen Joint Count (SJC) <= 1, C-Reactive Protein (CRP) <= 1 mg/dl and Patient's Global Assessment of Disease Activity (PtGADA) <= 10 mm.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 34.2 | 52.4 | 46.4

15. Secondary Outcome: Percentage of Subjects With Clinical Disease Activity Index (CDAI) <= 2.8 at Week 104 in RA0055 Period 2
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm). 28 joints are examined where a lower score indicates less disease activity.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 43.0 | 55.6 | 52.4

16. Secondary Outcome: Percentage of Subjects With Simplified Disease Activity Index (SDAI) <= 3.3 at Week 104 in RA0055 Period 2
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm) and C-Reactive Protein (CRP in mg/L). 28 joints are examined where a lower score indicates less disease activity.
  The SDAI score ranges from 0 to 86, with a negative value in SDAI change from Baseline indicating an improvement from Baseline.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 41.8 | 57.1 | 53.6

17. Secondary Outcome: Percentage of Subjects With Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28[ESR]) < 2.6 at Week 104 in RA0055 Period 2
Description: as for outcome 2
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 44.3 | 63.5 | 52.4

18. Secondary Outcome: Percentage of Subjects Meeting the 2011 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Remission Criteria Simplified for Clinical Practice at Week 104 in RA0055 Period 2
Description: The 2011 ACR/EULAR remission criteria simplified for clinical practice is defined as:
  Tender Joint Count (TJC) <= 1, Swollen Joint Count (SJC) <= 1 and Patient's Global Assessment of Disease Activity (PtGADA) <= 10 mm.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 35.4 | 52.4 | 50.0

19. Secondary Outcome: Percentage of Subjects Achieving a Good or Moderate European League Against Rheumatism (EULAR) Response at Week 104 in RA0055 Period 2
Description: Good response is defined as:
  DAS28[ESR] <= 3.2 and decrease from Baseline by >1.2;
  moderate response is defined as achievement of one of the following:
  * DAS28[ESR] <= 3.2 and decrease from Baseline > 0.6 and ≤ 1.2
  * DAS28[ESR] > 3.2 and ≤ 5.1 and decrease from Baseline > 0.6
  * DAS28[ESR] > 5.1 and decrease from Baseline >1.2.
  LOCF= Last Observation Carried Forward
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: FAS2 with LOCF. FAS2 did not include subjects who had received PBO+MTX in Period1 as this was not part of the study objectives for the Period2 efficacy analyses
  1 subject in the CZP+MTX/CZP Q2W+MTX and 1 in the CZP+MTX/PBO+MTX arm had post Week 52 assessments, but weren´t dosed in Period2. They are included in the FAS2, but excluded from the SS2
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 88.6 | 98.4 | 94.0

20. Secondary Outcome: Change From Baseline in Previous Study RA0055 Period 1 in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) to Week 104 in RA0055 Period 2
Description: DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x PtGADA, where 28 joints are examined and a lower score indicates less disease activity. DAS28[ESR] ranges from 0-10 with higher values representing higher disease activity.
  A negative value in DAS28[ESR] change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | -3.436 (1.711) | -4.252 (1.275) | -3.901 (1.546)

21. Secondary Outcome: Change From Week 52 in Previous Study RA0055 Period 1 in Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) to Week 104 in RA0055 Period 2
Description: as for outcome 20
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | 1.145 (1.372) | 0.414 (1.033) | 0.511 (1.215)

22. Secondary Outcome: Change From Baseline in Previous Study RA0055 Period 1 in Clinical Disease Activity Index (CDAI) to Week 104 in RA0055 Period 2
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm). 28 joints are examined. CDAI ranges from 0-76 with lower scores indicating less disease activity and higher scores indicating higher disease activity.
  A negative value in CDAI change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | -30.7 (16.4) | -37.2 (12.1) | -32.6 (15.5)

23. Secondary Outcome: Change From Week 52 in Previous Study RA0055 Period 1 in Clinical Disease Activity Index (CDAI) to Week 104 in RA0055 Period 2
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm). 28 joints are examined. CDAI ranges from 0-76 with lower scores indicating less disease activity and higher scores indicating higher disease activity.A negative value in CDAI change from Baseline indicates an improvement from Baseline.
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | 6.0 (10.4) | 1.7 (5.9) | 2.5 (7.9)

24. Secondary Outcome: Change From Baseline in Previous Study RA0055 Period 1 in Simplified Disease Activity Index (SDAI) to Week 104 in RA0055 Period 2
Description: as for outcome 16
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | -31.6 (17.4) | -39.1 (13.5) | -34.3 (16.8)

25. Secondary Outcome: Change From Week 52 in Previous Study RA0055 Period 1 in Simplified Disease Activity Index (SDAI) to Week 104 in RA0055 Period 2
Description: as for outcome 16
Time Frame: From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | 6.5 (10.9) | 1.7 (6.0) | 2.6 (7.8)

26. Secondary Outcome: Percentage of Subjects With a Health Assessment Questionnaire- Disability Index (HAQ-DI) ≤ 0.5 at Week 104 in RA0055 Period 2
Description: Normative physical function is defined as HAQ-DI score <= 0.5. The domains of the HAQ-DI are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities.
  The total score ranges from 0 to 3 with lower scores meaning lower disability.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 49.4 | 63.5 | 61.9

27. Secondary Outcome: Percentage of Subjects With Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) <= 3.2 at Week 104 in RA0055 Period 2
Description: as for outcome 2
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 59.5 | 73.8 | 65.5

28. Secondary Outcome: Time to Flare From Week 52 in RA0055 Period 1 to Week 104 in RA0055 Period 2
Description: Time to flare, defined as an increase of DAS28[ESR] >= 0.6 above Week 52 DAS28[ESR] level, having a DAS28[ESR] >= 3.2 and judged by the Investigator as due to RA and all three criteria confirmed at an additional visit two weeks thereafter, from Week 52 onwards.
  Data not available as > 75% of the participants failed to meet flare criteria.
Time Frame: Week 104 in RA0055 Period 2
Population: FAS2 did not include subjects who had received PBO + MTX in Period 1 as this was not part of the study objectives for the Period 2 efficacy analyses.
  1 subject in the CZP+MTX/CZP Q2W+MTX and 1 in the CZP+MTX/PBO+MTX arm had post Week 52 assessments, but weren´t dosed in Period 2. They are included in the FAS2, but excluded from the SS2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
days | NA (NA) — Data not available as > 75% of the participants failed to meet flare criteria. | NA (NA) — Data not available as > 75% of the participants failed to meet flare criteria. | NA (NA) — Data not available as > 75% of the participants failed to meet flare criteria.

29. Secondary Outcome: Change From Baseline in Previous Study RA0055 Period 1 in the Bristol Rheumatoid Arthritis Fatigue- Multidimensional Questionnaire (BRAF-MDQ) Total Score to Week 104 in RA0055 Period 2
Description: BRAF-MDQ total score ranges from 0 to 70 (with higher scores indicating worse fatigue), whereas the score for each dimension is different due to the varied number of questions (0 -22 for physical, 0- 21 for living, 0- 15 for cognition, and 0- 12 for emotion). A negative value in BRAF-MDQ change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) in RA0055 Period 1 to Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | -15.9 (16.7) | -21.6 (16.9) | -20.7 (17.3)

30. Secondary Outcome: Number of Work Days Missed (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: Number of work days missed in the last month for employed subjects.
Time Frame: Week 104 in RA0055 Period 2
Population: FAS2 with LOCF. FAS2 did not include subjects who had received PBO + MTX in Period1 as this was not part of the study objectives for the Period2 efficacy analyses
  1 subject in the CZP+MTX/CZP Q2W+MTX and 1 in the CZP+MTX/PBO+MTX arm had post Week 52 assessments, but weren´t dosed in Period2. They are included in the FAS2, but excluded from the SS2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
days | 0.5 (1.46) | 0.2 (0.89) | 0.3 (0.86)

31. Secondary Outcome: Number of Work Days With Reduced Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: Number of work days with reduced productivity in the last month for employed subjects.
  Only the employed subjects were analyzed.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 52 | 79 | 51
days | 1.5 (4.88) | 0.6 (2.01) | 0.8 (2.29)

32. Secondary Outcome: Interference With Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: The Arthritis interference in the last month with work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference) for employed subjects.
  Only the employed subjects were analyzed.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 52 | 79 | 51
units on a scale | 2.3 (2.84) | 0.9 (1.60) | 1.2 (2.19)

33. Secondary Outcome: Number of Days With no Household Work (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: Number of days with no household work in the last month.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
days | 1.4 (3.35) | 0.7 (2.29) | 0.8 (2.76)

34. Secondary Outcome: Number of Days With Reduced Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: Number of days with reduced household work productivity in the last month.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
days | 1.8 (4.49) | 0.9 (3.01) | 1.0 (3.37)

35. Secondary Outcome: Number of Days With Hired Outside Help (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: Number of days with hired outside help days in the last month.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
days | 0.3 (0.98) | 0.3 (2.70) | 0.1 (0.45)

36. Secondary Outcome: Number of Days Missed of Family/Social/Leisure Activities (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: Number of days missed of family/social/leisure activities in the last month.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
days | 1.2 (3.36) | 0.2 (1.80) | 0.2 (0.75)

37. Secondary Outcome: Interference With Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 104 in RA0055 Period 2
Description: The Arthritis interference in the last month with household productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference).
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
units on a scale | 2.0 (2.63) | 1.0 (1.53) | 1.1 (1.95)

38. Secondary Outcome: Percentage of Subjects Achieving Low Disease Activity (LDA) at Week 104 in RA0055 Period 2
Description: LDA is defined as achieving a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) <= 3.2.
  DAS28 values range from 2.0 to 10.0 with a higher value indicating a higher disease activity.
Time Frame: Week 104 in RA0055 Period 2
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | CZP+MTX / PBO+MTX (Full Analysis Set) | CZP+MTX / CZP Q4W+MTX (Full Analysis Set) | CZP+MTX / CZP Q2W+MTX (Full Analysis Set)
Number analyzed (Participants) | 79 | 126 | 84
percentage of subjects | 68.4 | 74.6 | 70.2

ADVERSE EVENTS:
Time Frame: Adverse events for Period 2 were collected from the date of the Week 52 study medication up to 70 days after the last (most recent) Certolizumab pegol (CZP) or Placebo (PBO) dose
Description: For the safety results, the main comparisons of interest are across the 3 CZP re-randomized groups; the PBO+MTX/PBO+MTX group is included for completeness.
  For subjects induced/ re-induced with CZP due to flare, only AEs up to the time of induction/re-induction with CZP are included. Note that 3 SAEs occurred after induction/ re-induction.
Arm/Group | PBO+MTX / PBO+MTX | CZP+MTX / PBO+MTX | CZP+MTX / CZP Q4W+MTX | CZP+MTX / CZP Q2W+MTX
Serious Adverse Events (participants affected / at risk) | 4/66 | 6/81 | 9/127 | 4/83
Other Adverse Events (participants affected / at risk) | 3/66 | 13/81 | 32/127 | 13/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PBO+MTX / PBO+MTX (N=66) | CZP+MTX / PBO+MTX (N=81) | CZP+MTX / CZP Q4W+MTX (N=127) | CZP+MTX / CZP Q2W+MTX (N=83)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Latent tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myxoid liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0/3 (0) | 0/10 (0) | 0/3 (0) | 1/7 (1) — Only subjects who were induced/re-induced with CZP in Period 2 due to flare are included
Bronchial carcinoma (Respiratory, thoracic and mediastinal disorders) | 0/3 (0) | 1/10 (1) | 0/3 (0) | 0/7 (0) — Only subjects who were induced/re-induced with CZP in Period 2 due to flare are included
Depression (Psychiatric disorders) | 0/3 (0) | 1/10 (1) | 0/3 (0) | 0/7 (0) — Only subjects who were induced/re-induced with CZP in Period 2 due to flare are included
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBO+MTX / PBO+MTX (N=66) | CZP+MTX / PBO+MTX (N=81) | CZP+MTX / CZP Q4W+MTX (N=127) | CZP+MTX / CZP Q2W+MTX (N=83)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 4 (4) | 5 (9)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 13 (15) | 4 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 5 (5) | 2 (2)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 8 (8) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days